CLINICAL TRIAL: NCT01949298
Title: Immediate vs Delayed Loading of Two Implants Supporting a Locator Retained Mandibular Overdenture - A Randomized Controlled Study
Brief Title: Immediate vs Delayed Loading of Two Implants Supporting a Mandibular Over Denture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: Dentsply Astra tech (Unknown)
Responsible Party: Principal Investigator, Gian Schincaglia, Clinical Associate Professor, UConn Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IE-10-305-3
Record Dates: First submitted 2013-09-19; First posted 2013-09-24 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Implant Survival Using Immediate Loading Protocol
Keywords: immediate loading of dental implant; implant supported over denture

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate implant loading (Experimental): The test group had implant immediately loaded by means of a implant supported mandibular denture connected with locator abutment.
  Interventions: Procedure: dental implant placement
- Delayed implant loading group (Active Comparator): The control group had implant loaded after 3 months of submerged healing by means of a implant supported mandibular denture connected with locator abutment.
  Interventions: Procedure: dental implant placement

INTERVENTIONS:
Procedure: dental implant placement

SUMMARY:
Edentulous patients have to wait after extractions and again after surgical implant placement for healing to occur before the implants can be restored and patients can go back to normal function. This delay in loading of implants can be handicapping for the patient, esthetically and functionally. Hence this project was undertaken with the purpose of reducing this wait period and achieving early rehabilitation in these patients. The aim of the project is to compare immediate loading versus delayed loading of implant supported mandibular dentures.

ELIGIBILITY:
Inclusion Criteria:

* Males and females at least >=21y of age
* Provision of informed consent
* Totally edentulous arch requiring or wearing mandibular complete denture
* Tooth in implant sites must have been extracted at least 4 months before the implant placement.
* Adequate amount of bone support to insert a 8mm in length and 4mm in diameter implant without encroaching on vital structures. The amount of bone available should be such that after implant placement there should be minimum of 1mm lingual and buccal bone
* Implant insertion torque >=20Ncm
* No need for bone augmentation procedures

Exclusion Criteria:

* Conditions or circumstances as evaluated by the investigator, which would prevent completion of study participation.
* Conditions requiring chronic routine use of antibiotics or requiring prolonged use of steroids.
* History of leukocyte dysfunction or deficiencies, bleeding disorders, neoplastic disease requiring radiation or chemotherapy, metabolic bone disorder, uncontrolled endocrine disorders, HIV infection
* Use of investigational drugs or devices within 30 days of study period,
* Alcoholism or drug abuse and heavy smokers > 10 cigarettes a day.
* Local factors such as

  * untreated periodontitis,
  * erosive lichen planus,
  * local irradiation history,
  * osseous lesion,
  * unhealed extraction socket,
  * intraoral infection,
  * lack of primary stability
  * inadequate oral hygiene
* Simultaneous participation in another clinical study

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2010-07; Primary Completion 2014-01 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Radiographic bone level change around the implants | 12 months

SECONDARY OUTCOMES:
Implant survival | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States

REFERENCES:
- [Background] Marzola R, Scotti R, Fazi G, Schincaglia GP. Immediate loading of two implants supporting a ball attachment-retained mandibular overdenture: a prospective clinical study. Clin Implant Dent Relat Res. 2007 Sep;9(3):136-43. doi: 10.1111/j.1708-8208.2007.00051.x. PMID 17716257
- [Derived] Schincaglia GP, Rubin S, Thacker S, Dhingra A, Trombelli L, Ioannidou E. Marginal Bone Response Around Immediate- and Delayed-Loading Implants Supporting a Locator-Retained Mandibular Overdenture: A Randomized Controlled Study. Int J Oral Maxillofac Implants. 2016 Mar-Apr;31(2):448-58. doi: 10.11607/jomi.4118. PMID 27004292